CLINICAL TRIAL: NCT01004757
Title: Improvement of Myocardial Function and Metabolic Syndrome in Type 2 Diabetes Patients by a Low Glycemic and Insulinemic Diet (LOGI®) Compared to the Traditional Low Fat Diet - a Prospective Parallel Group/Cross Over Study
Brief Title: Effects of Low Versus High Carbohydrate Diet During Rehabilitation on Cardiovascular Function and Metabolism in Type 2 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Munich Municipal Hospital (Other)
Collaborators: Stately Pension System (LVA) Baden-Wuertemberg (Unknown); Ueberruh Rehabilitation Clinic, Isny, Baden-Wuertemberg (Unknown)
Responsible Party: Prof. Dr. Helene von Bibra, Munich Municipal Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: LOGILoFaReha
Record Dates: First submitted 2009-10-29; First posted 2009-10-30 (Estimated); Last update posted 2009-10-30 (Estimated); Status verified 2009-10

CONDITIONS: Type 2 Diabetes Mellitus; Overweight
Keywords: diastolic function; postmeal glucose; insulin resistance; low carb diet; type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Overweight; Insulin Resistance | interventions — Diet, Fat-Restricted

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LOGI diet (Active Comparator): diet based on 25% low glycemic index carbohydrates, 30% protein and 45% fat combined with heart rate controlled, aerobic exercise
  Interventions: Other: LOGI diet
- Low Fat diet (Active Comparator): cross over design of three weeks Low Fat diet followed by two weeks LOGI diet always combined with heart rate controlled aerobic exercise
  Interventions: Other: Low Fat diet

INTERVENTIONS:
Other: LOGI diet — diet based on 25% low glycemic index carbohydrates, 30% protein and 45% fat combined with heart rate controlled aerobic exercise for three weeks
  Arms: LOGI diet
Other: Low Fat diet — traditional low fat diet based on 55% mixed glycemic index carbohydrates, 20% protein and 25% fat for three weeks followed by LOGI diet for two weeks, always combined with heart rate controlled aerobic exercise
  Arms: Low Fat diet

SUMMARY:
Compared to the traditional low fat diet for overweight patients with type 2 diabetes, recent evidence shows that low carbohydrate/high protein diets lower triglycerides and postprandial glucose levels more effectively. However, it is not known, whether this diet can also improve the subclinically impaired myocardial function in type 2 diabetes. This prospective parallel group and cross over design study compares the effects of a low glycemic and insulinemic diet (LOGI®) with an isocaloric traditional low fat diet during a three weeks rehabilitation programme with aerobic exercise for overweight type 2 diabetes patients testing the hypothesis, that the low carbohydrate diet improves myocardial function and insulin resistance.

DETAILED DESCRIPTION:
This is a single center, short term therapy controlled and prospective study with blinded analyses of the ultrasound data in 41 patients with type 2 diabetes either on dietary control or oral antidiabetic medication. After recruitment and informed consent, patients are randomized to two treatment arms matched for age and concomittant antidiabetic and cardiovascular medication In one treatment arm, the diet is based on the LOGI components: 25% low glycemic index carbohydrates, 30% protein, 45% fat, taken for 3 weeks combined with aerobic exercise, while in the other treatment arm, the isocaloric traditional low fat diet is based on 55% mixed glycemic index carbohydrates, 20 % protein and 25% fat taken for three weeks and combined with the same aerobic exercise protocoll but followed by a two weeks period with LOGI diet and maintained exercise. In both treatment arms, antidiabetic and antihypertensive medication are maintained and/or adapted as necessary and recorded.

All patients receive life style instructions and are updated in their skills of measuring quantity of foods and designing diet plans based on food groups. Laboratory, clinical and ultrasound investigations are performed before and at the end of the three weeks programme and, in the cross over group, also at the end of the subsequent diet programme.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes
* oral antidiabetic medication or dietary control
* overweight

Exclusion Criteria:

* coronary artery disease

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2008-02; Primary Completion 2009-12 (Estimated); Study Completion 2010-02 (Estimated)

PRIMARY OUTCOMES:
myocardial diastolic function | 2-3 weeks treatment period

SECONDARY OUTCOMES:
triglycerides, insulin resistance | 2-3 weeks treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Helene von Bibra, MD, PhD, Principal Investigator — Munich Academic Teaching Hospital Bogenhausen
Locations (1):
- Staedt. Klinikum Muenchen-Bogenhausen, Munich, Bavaria, Germany

REFERENCES:
- [Background] Hession M, Rolland C, Kulkarni U, Wise A, Broom J. Systematic review of randomized controlled trials of low-carbohydrate vs. low-fat/low-calorie diets in the management of obesity and its comorbidities. Obes Rev. 2009 Jan;10(1):36-50. doi: 10.1111/j.1467-789X.2008.00518.x. Epub 2008 Aug 11. PMID 18700873
- [Background] Gannon MC, Nuttall FQ. Effect of a high-protein, low-carbohydrate diet on blood glucose control in people with type 2 diabetes. Diabetes. 2004 Sep;53(9):2375-82. doi: 10.2337/diabetes.53.9.2375. PMID 15331548
- [Background] Yu CM, Sanderson JE, Marwick TH, Oh JK. Tissue Doppler imaging a new prognosticator for cardiovascular diseases. J Am Coll Cardiol. 2007 May 15;49(19):1903-14. doi: 10.1016/j.jacc.2007.01.078. Epub 2007 Apr 30. PMID 17498573
- [Background] Von Bibra H, Thrainsdottir IS, Hansen A, Dounis V, Malmberg K, Ryden L. Tissue Doppler imaging for the detection and quantitation of myocardial dysfunction in patients with type 2 diabetes mellitus. Diab Vasc Dis Res. 2005 Feb;2(1):24-30. doi: 10.3132/dvdr.2005.002. PMID 16305069
- [Background] von Bibra H, Hansen A, Dounis V, Bystedt T, Malmberg K, Ryden L. Augmented metabolic control improves myocardial diastolic function and perfusion in patients with non-insulin dependent diabetes. Heart. 2004 Dec;90(12):1483-4. doi: 10.1136/hrt.2003.020842. No abstract available. PMID 15547039